CLINICAL TRIAL: NCT02612233
Title: Pain Management in Osteoarthritis Using the Centrally Acting Analgesics Duloxetine and Pregabalin
Acronym: DUPRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: Rosetrees Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11.0126; 2011-003803-39 (EudraCT Number)
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Hand Osteoarthritis
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Pregabalin; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pregabalin (Active Comparator): Pregabalin 150mg ON week 1 increased to Pregabalin 300mg ON weeks 2-11 then decrease to Pregabalin 150mg ON week 12 then STOP
  Interventions: Drug: Pregabalin or Duloxetine or Placebo
- Duloxetine (Active Comparator): Duloxetine 30mg ON week 1 increase to Duloxetine 60mg weeks 2-11 then decrease to Duloxetine 30mg ON week 12 then STOP
  Interventions: Drug: Pregabalin or Duloxetine or Placebo
- Placebo (Placebo Comparator): 1 capsule ON week 1- increase to 2 capsules ON week 2-11 then decrease to 1 capsule ON week 12 then STOP.
  Interventions: Drug: Pregabalin or Duloxetine or Placebo

INTERVENTIONS:
Drug: Pregabalin or Duloxetine or Placebo — This is a randomized, double blind placebo controlled trial with a head-to-head comparison of duloxetine vs pregabalin vs placebo over-encapsulated to prevent unblinding of treatment arm
  Other Names: DUPRO Capsules

SUMMARY:
Osteoarthritis is the most common form of arthritis worldwide. Specifically, osteoarthritis of the hands affects millions of people and is a major cause of hand disability and pain. Despite this, there are currently no treatments that delay or halt the development of osteoarthritis. Pain is one of the major symptoms of osteoarthritis and pain management is an important factor to consider in the treatment of this condition. Treatments for pain in osteoarthritis consists of local injections, anti-inflammatory gels or painkillers such as paracetamol. However, most people with osteoarthritis still have pain despite these treatments.

DETAILED DESCRIPTION:
Recent scientific studies have suggested that people with hand osteoarthritis not only feel pain in their hand joints, they also appear to have increased signals in their brain pain processing pathways. At St George's, University of London, the investigators have been conducting studies to find out which brain regions are activated in subjects with hand osteoarthritis. The investigators have found that certain brain regions (thalamus, insula, cingulate and somatosensory cortex) are activated during painful tasks in patients with hand osteoarthritis but not in healthy people. In this study the investigators will establish whether drugs that inhibit pain processing pathways in the brain can help. Patients who are still having pain despite their usual painkillers will be randomly divided into 3 groups: one group will receive a placebo, the other 2 groups will receive one of two different drugs, duloxetine or pregabalin. Participants will be assessed using questionnaires and a brain scan (functional MRI) before and after 13 weeks of taking the tablets. This study will help us to understand the ways in which people feel pain in osteoarthritis. If our trial proves successful,drugs that dampen central pain pathways could be used in combination with local pain-relieving drugs to improve treatment and reduce disability in patients with hand osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Participants fulfilling the American College of Rheumatology (ACR) criteria for the diagnosis of hand osteoarthritis
* Participants with hand osteoarthritis presenting to rheumatology outpatient clinics and primary care.
* Participants will be right or left handed
* Male or female
* Age between 40 and 75
* Participants will be on usual care for hand osteoarthritis including paracetamol and/or non-steroidal anti-inflammatory drugs

Exclusion Criteria:

* Participants with other rheumatological diagnoses e.g. rheumatoid arthritis
* Current or planned pregnancy
* Contraindications to duloxetine or pregabalin
* History of depression
* Recent surgery
* Previous use of duloxetine and/or pregabalin

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Australian/Canadian Hand Osteoarthritis Index score (AUSCAN) | 12 weeks
  The AUSCAN measures pain and hand function. Differences between baseline AUSCAN and after treatment will be recorded for each participant to assess for improvement in AUSCAN pain and function score after the trial intervention.

SECONDARY OUTCOMES:
Brain magnetic resonance imaging (MRI) | Baseline and 12 weeks after treatment
  Changes between baseline MRI and post-treatment after 12 weeks of intervention will be measured using functional neuroimaging to assess pain center activation before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Sofat, MBBS, PhD, Principal Investigator — St George's, University of London
Locations (1):
- Hotung Centre for Musculoskeletal Diseases, London, United Kingdom